CLINICAL TRIAL: NCT02507817
Title: The Correlation Between LIF Levels in Cord Blood to Maternal Blood in Women Treated With Mg During Labor
Brief Title: Correlation Between LIF (Leukemia Inhibitory Factor ) Levels in Cord and Maternal Blood in Women Treated With Mg
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0604-14-RMB CTIL
Record Dates: First submitted 2015-06-25; First posted 2015-07-24 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: LIF LEVELS IN CORD BLOOD AND MATERNAL BLOOD DURING LABOR
Keywords: LIF,Magnesium Sulphate
MeSH Terms: interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples without DNA

GROUPS / COHORTS (4):
- 31-32 with Mg for neuroprotection: Women in 31-32 weeks gestation that where treated with Magnesium Sulphate for neuroprotection.
  blood sample and tissue sample (placenta).
  Interventions: Other: blood sample and tissue sample
- 33-34 without Mg for neuroprotection: Women in 33-34 weeks gestation that per protocol are not entitled for treatment with Magnesium Sulphate for neuroprotection.
  blood sample and tissue sample (placenta).
  Interventions: Other: blood sample and tissue sample
- PET with Mg after 34 weeks: Women that had severe preeclamsia and where treated with Magnesium Sulphate for seizure prophylaxis and delivere after 34 weeks of gestation.
  blood sample and tissue sample (placenta).
  Interventions: Other: blood sample and tissue sample
- control: Low risk pregnanacies in similar weeks to group 3 that did not require any special teatment and delivered after 34 weeks of gestation.
  blood sample and tissue sample (placenta).
  Interventions: Other: blood sample and tissue sample

INTERVENTIONS:
Other: blood sample and tissue sample — Maternal LIF levels prior and after delivery.After birth and disconnection of the cord, we also will take a blood sample from the umbilical cord (5cc) for cytokine ELISA testing.
  A small sample of the placenta will be examined in order to assess the level of ACTH protein

SUMMARY:
During embryonic development, there are several cytokines such as: LIF (Leukemia inhibitory factor), ciliary neurotrophic factor (CNTF), epidermal growth factor family (EGF), neuregulin 1 (NRG1) and transforming growth factor β (TGFβ) that were found are associated with neurogenesis and differentiation of brain cells.

LIF is a cytokine that is essential for the development of the central nervous system, and has recently been shown in rats that maternal LIF stimulates placental ACTH (adrenocorticotropic hormone) that in turn promotes secretion of fetal LIF from nRBC (nucleated red blood cell ), which in turn promotes brain development of the fetus In other studies on rats a theory was proposed that LPS (lipopolysaccharide) and infection during pregnancy influence the normal development of the brain and may cause brain damage by altering placental ACTH thank in turn alters LIF secretion in the embryo which could be the cause of brain damage.

Our hypothesis is that by treating the mother with Magnesium Sulphate we can protect the embryo's brain in one of two ways:

1. Altering Placental ACTH
2. Altering the number of receptors for LIF in the brain Women who are at risk for preterm labor prior to 32 weeks of gestation are treated with Magnesium Sulphate for neuroprotection, randomized controlled studies showed that if these women are treated in the 24 hours prior to labor with magnesium sulphate the risk for cerebral palsy and other severe motor problems are decreased.

The mechanism for this decrease is unknown and that is the purpose of our study.

The purpose of our research is to examine maternal LIF levels prior to birth and Maternal and cord levels after delivery and to see if levels are different if the mother was treated with Magnesium Sulphate. We will also check the placental ACTH level

DETAILED DESCRIPTION:
During embryonic development, there are several cytokines such as: LIF (Leukemia inhibitory factor), ciliary neurotrophic factor (CNTF), epidermal growth factor family (EGF), neuregulin 1 (NRG1) and transforming growth factor β (TGFβ) that were found are associated with neurogenesis and differentiation of brain cells.

LIF is a cytokine that is essential for the development of the central nervous system, and has recently been shown in rats that maternal LIF stimulates placental ACTH (adrenocorticotropic hormone) that in turn promotes secretion of fetal LIF from nRBC (nucleated red blood cell ), which in turn promotes brain development of the fetus In other studies on rats a theory was proposed that LPS (lipopolysaccharide) and infection during pregnancy influence the normal development of the brain and may cause brain damage by altering placental ACTH thank in turn alters LIF secretion in the embryo which could be the cause of brain damage.

Our hypothesis is that by treating the mother with Magnesium Sulphate we can protect the embryo's brain in one of two ways:

1. Altering Placental ACTH
2. Altering the number of receptors for LIF in the brain Women who are at risk for preterm labor prior to 32 weeks of gestation are treated with Magnesium Sulphate for neuroprotection, randomized controlled studies showed that if these women are treated in the 24 hours prior to labor with magnesium sulphate the risk for cerebral palsy and other severe motor problems are decreased.

The mechanism for this decrease is unknown and that is the purpose of our study.

The purpose of our research is to examine maternal LIF levels prior to birth and Maternal and cord levels after delivery and to see if levels are different if the mother was treated with Magnesium Sulphate. We will also check the placental ACTH level .

ELIGIBILITY:
Inclusion Criteria:

1. Women in 31-32 weeks gestation that where treated with Magnesium Sulphate for neuroprotection.
2. Women in 33-34 weeks gestation that per protocol are not entitled for treatment with Magnesium Sulphate for neuroprotection.
3. Women that had severe preeclampsia and where treated with Magnesium Sulphate for seizure prophylaxis and delivered after 34 weeks of gestation.
4. Low risk pregnancies in similar weeks to group 3 that did not require any special treatment and delivered after 34 weeks of gestation

Exclusion Criteria:

- Women who do not agree known genetic diseases or fetal abnormality

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Women in 31-32 weeks gestation that where treated with Magnesium Sulphate for neuroprotection.
  2. Women in 33-34 weeks gestation that per protocol are not entitled for treatment with Magnesium Sulphate for neuroprotection.
  3. Women that had severe preeclampsia and where treated with Magnesium Sulphate for seizure prophylaxis and delivered after 34 weeks of gestation.
  4. Low risk pregnanacies in similar weeks to group 3 that did not require any special teatment and delivered after 34 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between LIF Levels in women who where treated with Mg and women who where not (maternal LIF levels prior to birth and Maternal and cord levels after delivery) | 2 years